CLINICAL TRIAL: NCT00928785
Title: A Randomised, Comparative, Multicentre Clinical Trial of the Immunogenicity and Safety of Tdap-IPV Vaccine and a Tetanus Monovalent Vaccine in Healthy Adults 18 Years of Age and Older
Brief Title: Study Comparing a Tdap-IPV Combined Vaccine With a Tetanus Monovalent Vaccine in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RPV02C
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Tetanus Vaccine; Tdap-IPV vaccine
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- REPEVAX (Experimental)
  Interventions: Biological: REPEVAX
- Monovalent tetanus vaccine (Active Comparator)
  Interventions: Biological: Monovalent Tetanus vaccine

INTERVENTIONS:
Biological: REPEVAX — 1 dose of 0.5 mL at Day 0
  Arms: REPEVAX
Biological: Monovalent Tetanus vaccine — 1 dose of 0.5 mL at Day 0
  Arms: Monovalent tetanus vaccine

SUMMARY:
The purpose of this study is to demonstrate that a combined adult Tdap-IPV vaccine (REPEVAX®) will provide similar rapid antibody responses against tetanus toxoid as a tetanus toxoid vaccine alone in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥18 years
* Last booster with a T-containing vaccine received 5 to 10 years prior to the administration of the study vaccine (documented by written evidence)
* Subject with vaccination history of a primary immunisation with a tetanus, diphtheria and poliomyelitis containing vaccine as recommended in the local vaccination calendar
* Negative urine pregnancy test for female subjects of child-bearing potential. A female subject who is of reproductive potential must agree to remain abstinent or use (or have her partner use) acceptable methods of birth control during the study period
* Subject having signed the informed consent form prior to participation in the study

Exclusion Criteria:

* Acute severe illness or fever (>=38.0°C) within the last 3 days
* Hypersensitivity or known allergy to one of the components of one of the study vaccines (including formaldehyde, streptomycin, neomycin, polymyxin B, or glutaraldehyde)
* Anaphylactic or other allergic reactions to a previous dose of a vaccine containing diphtheria or tetanus toxoids or poliomyelitis viruses or pertussis (acellular or whole cell)
* Guillain Barré syndrome or neuropathy of brachial plexus following a previous vaccination with a tetanus toxoid containing vaccine
* Known encephalopathy after receipt of a pertussis vaccine or neurological disorders after an injection with the same antigens
* Progressive or unstable neurological disorder, uncontrolled seizures or progressive encephalopathy not stabilized
* Known malignant disease, note:

  * subjects with prostate or breast cancer who are not on chemotherapeutic drugs (other than hormone blocking drugs),
  * subjects with skin cancer who are not receiving radiation therapy or chemotherapy, and
  * subjects with a history of other malignancies who have been disease-free for at least 5 years will be eligible for enrollment
* Immunosuppressive therapy:

  * High dose (≥ 20 mg/day prednisone equivalent) systemic (≥ 14 days) corticosteroid treatment daily or on alternate day within the last 28 days (inhaled corticosteroids allowed)
  * Chemotherapeutic agents used to treat cancer or other conditions
  * Treatments associated with organ or bone marrow transplantation
* Immune dysfunction caused by a medical condition, or any other cause (e.g., congenital immunodeficiency, human immunodeficiency virus (HIV) infection, organ or bone marrow transplantation, leukemia, lymphoma, Hodgkin's disease, multiple myeloma or generalized malignancy)
* Known severe thrombocytopenia or coagulation disorder contraindicating an intramuscular injection
* Administration of blood products including immunoglobulins within the last 90 days or planned before Visit 3
* Recent administration of a live vaccine (≤28 days) or an inactivated vaccine (≤14 days) or vaccination planned before Visit 3
* For female subjects, pregnancy (positive pregnancy test before first blood sample) or breast-feeding through Visit 3
* Planned participation in another clinical study during the present study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Anti-tetanus seroprotection rate (defined as the percentage of subjects with anti-tetanus antibody titre (ELISA) ≥ 0.1 IU/mL) | 10 days

SECONDARY OUTCOMES:
Geometric Mean Titre (GMT) for tetanus antibodies in both groups | Day 0, Day 1 and Day 28
The anti-tetanus seroprotection rate (antibody titre ≥ 0.1 IU/mL in ELISA) | Day 28
Percentage of subjects with immediate reactions, solicited injection-site reactions, systemic reactions and unsolicited adverse events | D0 to Day 7
Percentage of subjects with serious adverse events | D0 to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (9):
- France (4):
  - Hôpital Gabriel Montpied - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital St Eloi, Montpellier
  - Groupe Hospitalier Cochin - Saint-Vincent de Paul, Paris
  - Hôpital Bichat Claude Bernard, Paris
- Germany (5):
  - Heilbronn
  - Künzig
  - Nettersheim
  - Offenbach
  - Reichenbach/Vogtland

REFERENCES:
- [Derived] Laurichesse H, Zimmermann U, Galtier F, Launay O, Duval X, Richard P, Sadorge C, Soubeyrand B. Immunogenicity and safety results from a randomized multicenter trial comparing a Tdap-IPV vaccine (REPEVAX(R)) and a tetanus monovalent vaccine in healthy adults: new considerations for the management of patients with tetanus-prone injuries. Hum Vaccin Immunother. 2012 Dec 1;8(12):1875-81. doi: 10.4161/hv.22083. Epub 2012 Oct 2. PMID 23032160